CLINICAL TRIAL: NCT07315789
Title: Effects of a High-intensity Interval Strength Training Programme in Institutionalized Older Adults With Sarcopenia: a Randomized Clinical Trial.
Brief Title: Effects of a Strength Training Programme in Institutionalized Older Adults With Sarcopenia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Jesús Zapata Linares, Clinical professor, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02
Record Dates: First submitted 2025-12-10; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia in Elderly; Institutionalized Older Adults; HIIT

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- This group includes institutionalized older adults aged 60 and over for treatment. (Experimental)
  Interventions: Other: High-intensity interval strength training: therapeutic exercise programme.
- This group includes institutionalized older adults aged 60 and over. (No Intervention)

INTERVENTIONS:
Other: High-intensity interval strength training: therapeutic exercise programme. — A 12-week high-intensity interval strenght training (HIITs) programme is developed with basic exercises adapted to the living environment of older people. Progress in the exercises over the twelve weeks is measured using the maximum weight that can be lifted in one repetition (1-RM), maximum heart rate (MHR) and the Borg scale.
  Arms: This group includes institutionalized older adults aged 60 and over for treatment.

SUMMARY:
Sarcopenia is one of the main problems in the elderly population. The concept of disease has evolved, as have its treatment strategies. Among these is high-intensity interval training (HIIT). This approach has been little studied in older adults with sarcopenia, especially in institutionalized older adults in nursing homes. So this will be the objective of the study. A randomised clinical trial is being conducted to analyse how these diagnostic criteria for sarcopenia evolve after the application of HIIT compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* older adults who have been institutionalized for at least one year
* older adults who are institutionalized with clinical suspicion of sarcopenia according to the Sarc-F questionnaire and muscle strength criteria
* older adults residing in the community of Extremadura.

Exclusion Criteria:

* present cognitive impairment (score <24 Mini-Mental State Examination)
* primary, serious, or chronic diseases that could explain the decrease in muscle strength and the other diagnostic variables of the participants
* diseases or physical disorders that hinder the assessment of the participants; -use of drugs that may affect muscle strength and mass.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Hand grip strenght | Thrice at the baseline: at the start, at 8 weeks and at 12 weeks.
  The researchers used the JAMAR dynamometer

SECONDARY OUTCOMES:
Muscular mass / appendicular skeletal mass (ASM) | Thrice at the baseline: at the start, at 8 weeks and at 12 weeks.
  The researchers used bioimpedance analysis with Tanita MC780-S MA Multifrequency.
Physical performance | Thrice at the baseline: at the start, at 8 weeks and at 12 weeks.
  The researchers used the scale: "Short Physical Performance Battery" (SPPB).
Physical performance 2 | Thrice at the baseline: at the start, at 8 weeks and at 12 weeks.
  The researchers used the test: "Timed Up and Go" (TUG).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Extremadura, Badajoz, Spain